CLINICAL TRIAL: NCT00052468
Title: A Multi-National Randomized Phase-III GCIG Intergroup-Study Comparing 1st-line Chemotherapy With Gemcitabine/Paclitaxel/Carboplatin vs Paclitaxel/Carboplatin In Previously Untreated Patients With Epithelial Ovarian Cancer FIGO Stages I-IV
Brief Title: Carboplatin/Paclitaxel +/-Gemcitabine in Treating Patients With Ovarian Epithelial or Fallopian Tube Cancer
Acronym: AGO-OVAR9
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AGO Study Group (Other)
Collaborators: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other); GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258429; AGO-OVAR9; NORDIC-AGO-OVAR-9; GERCOR-AGO-OVAR-9; EU-20241
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Paclitaxel; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TCG (Experimental): Paclitaxel 175 mg/m2 day 1, Carboplatin AUC 5 day 1, Gemcitabine 800 mg/m2 day 1 + 8, q 21 days / 6 - 10 courses
  Interventions: Drug: TCG
- TC (Active Comparator): Paclitaxel 175 mg/m2 day 1, Carboplatin AUC 5 day 1, q 21 days / 6 - 10 courses
  Interventions: Drug: TC

INTERVENTIONS:
Drug: TCG
  Other Names: Paclitaxel/Carboplatin/Gemcitabine
  Arms: TCG
Drug: TC
  Other Names: Paclitaxel/Carboplatin
  Arms: TC

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether carboplatin and paclitaxel combined with gemcitabine is more effective than carboplatin and paclitaxel alone in treating ovarian epithelial or fallopian tube cancer.

PURPOSE: This randomized phase III trial is studying carboplatin and paclitaxel combined with gemcitabine to see how well it works compared to paclitaxel and carboplatin alone in treating patients who have undergone surgery for ovarian epithelial or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare overall survival in patients with stage I-IV ovarian epithelial or fallopian tube cancer treated with adjuvant carboplatin and paclitaxel with or without gemcitabine.
* Compare response rates, progression-free survival, and duration of response in patients treated with these regimens.
* Compare toxic effects of these regimens in these patients.
* Compare quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, controlled, multicenter study. Patients are stratified according to FIGO stage (I-IIA vs IIB-IIIC and tumor no greater than 10 mm vs IIB-IIIC and tumor greater than 10 mm or IV), plan for interval surgical debulking (yes vs no), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive carboplatin IV over 30-60 minutes and paclitaxel IV over 3 hours on day 1 and gemcitabine IV over 30-60 minutes on days 1 and 8.
* Arm II: Patients receive carboplatin and paclitaxel as in arm I. Treatment in both arms repeats every 21 days for 6 to 10 courses in the absence of disease progression or unacceptable toxicity.

Some patients undergo interval debulking surgery.

Quality of life is assessed at baseline, after courses 3 and 6, and then at 3, 6, and 12 months after completion of study.

Patients are followed every 3 months for 2 years, every 6 months for up to 5 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,716 patients (858 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of one of the following:

  * Ovarian epithelial cancer

    * FIGO stage IA/B G3, IC-IV
  * Fallopian tube cancer
  * Extra-ovarian papillary serous tumor
* The following are ineligible:

  * Low malignant-potential ovarian tumors (borderline tumors)
  * Non-epithelial ovarian tumors
  * Mixed Mullerian tumors
* Must have had definitive surgery within the past 6 weeks
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 6 months

Hematopoietic

* WBC at least 3,000/mm^3 OR
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin greater than 10 mg/dL

Hepatic

* Bilirubin no greater than 2 times upper limit of normal

Renal

* Glomerular filtration rate at least 50 mL/min

Cardiovascular

* No congestive heart failure
* No myocardial infarction within the past 6 months
* No New York Heart Association class III or IV heart disease
* No prior atrial or ventricular arrhythmias

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior seizures or central nervous system disorder
* No prior severe hypersensitivity reaction to products containing Cremophor EL (e.g., cyclosporine or vitamin K)
* No known hypersensitivity to compounds chemically related to carboplatin, gemcitabine, or paclitaxel
* No preexisting motor or sensory neuropathy greater than grade 1
* No other malignancy within the past 5 years except:

  * Malignancies cured by surgery alone
  * Carcinoma in situ of the cervix
  * Adequately treated basal cell skin cancer
* No complete bowel obstruction
* No other concurrent severe medical condition that would preclude study participation
* No dementia or significantly altered mental status that would preclude study participation
* No concurrent severe active infection
* Geographically accessible for treatment and follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy except:

  * Hormone replacement therapy
  * Antiemetic steroids

Radiotherapy

* No prior radiotherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* Recovered from prior surgery

Other

* No other concurrent antineoplastic agents
* No other concurrent investigational drugs
* No other concurrent clinical trial enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1742 (Actual)
Dates: Start 2002-08; Primary Completion 2009-07 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Whole Study Period
  Survival time is calculated from the date of enrollment into the study until the date of death from any cause

SECONDARY OUTCOMES:
Progression Free Survival | Whole Study Period
  The progression-free survival is calculated for all patients from the date of enrollment until the date of first progressive disease or death, whichever occurs first

OTHER OUTCOMES:
Quality of Life | Whole Study Period

CONTACTS AND LOCATIONS:
Overall Officials: Andreas du Bois, MD, PhD, Study Chair — Dr. Horst-Schmidt-Kliniken; J. Herrstedt, Study Chair — Copenhagen County Herlev University Hospital; E. Pujade-Lauraine, MD, PhD, Study Chair — Hotel Dieu de Paris
Locations (17):
- Herlev Hospital - University Hospital of Copenhagen, Copenhagen, Denmark
- Hotel Dieu de Paris, Paris, France
- Germany (14):
  - Zentralkrankenhaus, Bremen
  - Evangelisches Krankenhaus, Düsseldorf
  - Universitaetsklinikum Essen, Essen
  - Staedtische Kliniken Frankfurt am Main - Hoechst, Frankfurt
  - Frauenklinik der MHH, Hanover
  - Vincentius Krankenhaus, Karlsruhe
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - Klinikum Grosshadern der Ludwig-Maximilians Universitaet Muenchen, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Klinik und Poliklinik fuer Frauenheilkunde und Geburtshilfe - Universitaetsklinikum Muenster, Münster
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaet Ulm, Ulm
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
- Norwegian Radium Hospital, Oslo, Norway

REFERENCES:
- [Result] du Bois A, Herrstedt J, Hardy-Bessard AC, Muller HH, Harter P, Kristensen G, Joly F, Huober J, Avall-Lundqvist E, Weber B, Kurzeder C, Jelic S, Pujade-Lauraine E, Burges A, Pfisterer J, Gropp M, Staehle A, Wimberger P, Jackisch C, Sehouli J. Phase III trial of carboplatin plus paclitaxel with or without gemcitabine in first-line treatment of epithelial ovarian cancer. J Clin Oncol. 2010 Sep 20;28(27):4162-9. doi: 10.1200/JCO.2009.27.4696. Epub 2010 Aug 23. PMID 20733132
- [Derived] Machelon V, Gaudin F, Camilleri-Broet S, Nasreddine S, Bouchet-Delbos L, Pujade-Lauraine E, Alexandre J, Gladieff L, Arenzana-Seisdedos F, Emilie D, Prevot S, Broet P, Balabanian K. CXCL12 expression by healthy and malignant ovarian epithelial cells. BMC Cancer. 2011 Mar 16;11:97. doi: 10.1186/1471-2407-11-97. PMID 21410972